CLINICAL TRIAL: NCT06393491
Title: Equine-assisted Therapy in the Management of Adolescent Patients With Severe Anorexia Nervosa: a Qualitative Study
Brief Title: Equine-assisted Therapy and Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: EQUINE-ASSISTED THERAPY
Record Dates: First submitted 2024-03-29; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-03

CONDITIONS: Anorexia Nervosa; Equine-Assisted Therapy
Keywords: Anorexia Nervosa; Equine-Assisted therapy; Animal-assisted therapy; Complementary therapy; Health Care
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Severe anorexia nervosa is a complex psychiatric pathology with limited therapeutic tools to reduce morbidity and mortality. Equine-assisted therapy could provide additional therapeutic benefits.

Objectives : The investigators aimed to explore the effects of equine assisted therapy on the experience of adolescents with severe anorexia nervosa.

Méthods : Using a qualitative approach based on Interpretative Phenomenological Analysis, the investigators conducted semi-structured interviews with nine participants who had taken part in equine-assisted therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* having participated in at least 2 equine-assisted therapy sessions
* being or having been hospitalised between 2016 and 2022 in the psychiatric hospitalisation unit of the Institut Mutualiste Montsouris (Paris)
* ICD 10 diagnosis F50.0/ F.50.1
* female gender
* age between 13 and 25
* fluent French
* consent (including parents if minor participant)

Exclusion Criteria:

* having been under the care of C. Lepy (resident) during hospitalisation at the Institut Mutualiste Montsouris (Paris)
* refusal to participate on the part of the participant or the holder of parental authority.

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female participants who were between 13 and 25 years old and had completed at least 2 sessions of equine-assisted therapy during a hospitalization for anorexia nervosa between 2016 and 2022 in the psychiatric hospitalisation unit of the Institut Mutualiste Montsouris (Paris)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Semi-structured face-to-face interviews of patients was carried out using the Interpretative Phenomenological Analysis (IPA) method. | Between November 2020 and May 2022, when participants had completed at least 2 sessions of equine-assisted therapy during a hospitalization for anorexia nervosa
  Interpretative Phenomenological Analysis (IPA) method : this method explores people's perception of experience and how they make sense of it.
  IPA is based on three epistemological foundations: phenomenology, hermeneutics and ideography. The phenomenological approach seeks to explore the participant's understanding of the world. Hermeneutics assumes the interpretive dimensions of the results, both in the participant's access to their own experience, and in the researcher's access to the participant's perception of the world.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie LETRANCHANT, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No